CLINICAL TRIAL: NCT03115320
Title: A Protocol for a Randomized, Two-Parallel-group Study to Compare the Efficacy of Testing LH Surge at Home Versus Medically Triggered Ovulation With hCG (Pregnyl®) in the Naturally Stimulated Cycle in the Frozen-thawed Embryo Transfer
Brief Title: Frozen-thawed Embryo Transfer in a Natural Cycle: hCG Triggering Versus LH Home Test
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: High cancellation rate in LH test group in interim analysis
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R16172M; 2016-003959-29 (EudraCT Number)
Record Dates: First submitted 2016-11-17; First posted 2017-04-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2020-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnyl (Human chorionic gonadotropin) (Experimental): In this group, patients have natural cycle in frozen-thawed embryo transfer and the ovulation is confirmed by administration of hCG (Pregnyl® 5000 IU). The day of transferring embryo is depending on the day of administration of hCG and the age of the embryo. The day zero day is defined by ovulation triggered by hCG.
  Interventions: Drug: Human chorionic gonadotropin
- Home ovulation test (Other): The patients randomized to the LH surge group perform the ovulation home test daily from the urine. Thus, the ovulation in this group is corfimed by the urine test. The day of transferring embryo is depending on the positive ovulation test and the age of the embryo. The day zero day is defined by positive ovulation test.
  Interventions: Other: Home ovulation test

INTERVENTIONS:
Drug: Human chorionic gonadotropin — Human chorionic gonadotropin (Pregnyl, 5000IU) is used in the medication group to confirme the ovulation.
  Other Names: Home ovulation test
  Arms: Pregnyl (Human chorionic gonadotropin)
Other: Home ovulation test — The ovulation in the natural menstrual cycle is confirmed by the home ovulation tests from the urine.
  Arms: Home ovulation test

SUMMARY:
The primary aim of this study is to find out if ovulation triggered with hCG provides any additional benefit in comparison to spontaneous LH surge measured with the LH surge home test when transferring frozen-thawed embryo in a natural cycle.

DETAILED DESCRIPTION:
The aim of this study is to find out the best method for the ovulation triggering. We study the live birth rates in the both groups.

ELIGIBILITY:
Inclusion Criteria:

* - Patient with IVF or ICSI cycle and therefore having frozen-thawed embryos
* Regular menstruation cycle
* Patient's willingness to participate in the study

Exclusion Criteria:

* - Irregular menstrual cycle demanding preparing endometrium with hormones for frozen-thawed embryo
* No frozen embryos after IVF cycle
* Allergy to Pregnyl® or some of its ingredients in the medication or other contraindications due to Pregnyl®

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Live birth rate | At possible delivery (about 40 weeks)
  Live birth rate

SECONDARY OUTCOMES:
Ongoing pregnancy rate | After two weeks
  Ongoing pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Helena Tinkanen, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland